CLINICAL TRIAL: NCT03265782
Title: Comparison Between the Effect of Oral Paracetamol Versus Oral Ibuprofen in the Treatment of Patent Ductus Arteriosus in Preterm and Low Birth Weight Infants
Brief Title: Paracetamol Versus Ibuprofen for PDA Closure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, pricipal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43214321
Record Dates: First submitted 2015-03-10; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Patent Ductus Arteriosus
Keywords: efficacy; safety; paracetamol; ibuprofen; PDA; preterms
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ibuprofen group (Experimental): treatment of pda with oral ibuprofen with a loading dose 10 mg/kg/ds in the first day followed by 5 mg/kg/ds in the second ant third days then a follow up echo is done
  Interventions: Drug: ibuprofen
- paracetamol group (Experimental): treatment of pda with oral paracetamol with dose of 15 mg/kg/ds every 6 hours for 3 days then a follow up echo is done
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: ibuprofen — drug was adminstred with a loading dose 10 mg/kg/day followed by 5 mg/kg/day in 2 doses with 24 hrs apart for 3 days
  Other Names: brufen
  Arms: ibuprofen group
Drug: paracetamol — drug was administred for 3 consequetive days in a dosev 15 mg/kg/dose every 6 hrs and follow up echo was done after 3 days
  Other Names: cetal
  Arms: paracetamol group

SUMMARY:
Comparison between the safety and efficacy of oral paracetamol and oral ibuprofen in treatment of Patent Ductus Arteriosus (PDA) in premature infants

DETAILED DESCRIPTION:
A pilot study through which we have studied efficacy and safety of oral paracetamol and oral ibuprofen in treatment of hemodyamically significant pda in preterm neonates. 30 preterm neonates were included in the study 15 per each group. echo was done in the beginning and during treatment with both drugs to follow up the closure of the duct.

Ibuprofen was given as 10 mg/kg/dose in the 1st day followed by 5 mg/kg/dose in the 2nd and 3rd days with follow up echo was done after finishing the course paracetamol was given as 15 mglkg/6 hrs for three days with follow up echo to check the ductal closure.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≤ 35 weeks
2. Aged 2-7 days with color Doppler echocardiographic evidence of PDA
3. Urine output more than 1 ml/kg/hr
4. Creatinine concentration level less than 1.8 mg/dl

Exclusion Criteria:

Neonates who have one or more of the following criteria were excluded from the study:

1. Congenital heart diseases of any type including

   * Pulmonary stenosis
   * Anomalus in pulmonary venous drainage
   * Ventricular septal defect
2. Major congenital anomalies as hydrops fetalis
3. Low platelets count (less than 60, 000/mm3)

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
closure of PDA | 6 days
  Echo confirmed closure

REFERENCES:
- [Derived] El-Farrash RA, El Shimy MS, El-Sakka AS, Ahmed MG, Abdel-Moez DG. Efficacy and safety of oral paracetamol versus oral ibuprofen for closure of patent ductus arteriosus in preterm infants: a randomized controlled trial. J Matern Fetal Neonatal Med. 2019 Nov;32(21):3647-3654. doi: 10.1080/14767058.2018.1470235. Epub 2018 May 9. PMID 29695206